CLINICAL TRIAL: NCT00202761
Title: Project:Intensive Habilitation (PIH) -a New Norwegian Multidisciplinary Program for Intensive Training for Children With Disabilities
Brief Title: Project:Intensive Habilitation (PIH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Principal Investigator, Sissel Ledang, Research administrator, Sorlandet Hospital HF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SSHF70339
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Functional training; preschool children; Gross Motor Functional Classification Level; Gross motor functional Measure test; Pediatric Evaluation of Disability Inventory; Parental Stress Index
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PIH (Experimental): Intensified training of children with CP. Functional training (motor, speech, executive function). Coaching of parents by psychologist, individually and in groups.
  Interventions: Behavioral: PIH

INTERVENTIONS:
Behavioral: PIH — Intensified training

SUMMARY:
The purpose of this study is to document that taking part in this program is beneficial for the child, its parents and local professionals.

The study hypothesis are:

Intensive training will speed up the childs motor, cognitive and social development.

Intensive habilitation will increase the childs family's empowerment Children having participated in this intensive habilitation will speed up their process of development further than children in the control group The cooperation between first and second line health service is strengthened by participation in the intensive habilitation program The professionals in the first line(community)in Norway that participates in this program increases their empowerment and motivation

ELIGIBILITY:
Inclusion Criteria:

About three years of age Cerebral Palsy Multidisciplinary diagnosed -

Exclusion Criteria:

Not have Pervasive Developmental Disorder (PDD) No Specific Speech and Language Disorders No Serious Sensory Defects -

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2004-03; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
PEDI | dec 2006

SECONDARY OUTCOMES:
PSI | Dec 2006

CONTACTS AND LOCATIONS:
Overall Officials: Jon Skranes, MD, PhD, Principal Investigator — Sorlandet Hospital HF
Locations (1):
- Sorlandet Hospital HF, Kristiansand, Norway

REFERENCES:
- See also: Page describing the intensive habilitation program, and the childrens habilitation department at Sorlandet Hospital, HF , Norway — http://www.habu.no